CLINICAL TRIAL: NCT02186067
Title: Developing an Integrated System Approach for the Management of Hypertension: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Waris Qidwai, Professor and Chairman Department of Family Medicine, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13102013FM
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
Keywords: Hypertension; Uncontrolled Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Referral System (Experimental): Referral System:
  Primary Level Secondary Level Tertiary Level
  Interventions: Other: Referral System
- Control (No Intervention): Usual/routine care will be provided to the patients

INTERVENTIONS:
Other: Referral System — Primary Level:
  Refer patients to secondary care centre if Patients has complicated hypertension (Patients with target organ damage, CVD, CKD or more the 3 drugs)
  Secondary Level:
  Community health center at Aga Khan University will serve as the secondary care center.
  Family physician will manage patients with CVD, CKD or more than 3 drugs.
  Tertiary care:
  Cardiologist at the Aga Khan University will manage secondary, resistant and difficult to treat hypertension.
  Behavioral: Other Interventions CME session by Cardiologist/Consultant Family Physician : At start , and at two months Community screening by Family physicians at the primary care center (open house) once in three months Patient group education session. Once in three months
  Arms: Referral System

SUMMARY:
Hypertension has become a public health concern worldwide due to its significant contribution to the global health burden and its role as a prominent risk factor for the development of a number of chronic diseases such as Cardiovascular diseases (CVD), the leading cause of mortality in Pakistan and Worldwide. According to WHO, about 7.5 million deaths worldwide is attributable to hypertension i.e. about 12.8% of the total of all deaths. This accounts for 57 million disability adjusted life years (DALYS) or 3.7% of total DALYS.

Studies suggest that hypertension is among the top five most common presenting complaints to private general practice clinics. Therefore, primary care physicians/Family physicians are the first line service providers and; thus it is important to manage hypertensive patients early, through lifestyle and treatment interventions that may prevent the complications such as development of CVDs etc.

DETAILED DESCRIPTION:
To the best of authors' knowledge limited evidence is available from Pakistan on management of hypertension through an integrated approach. Therefore, the aim of the trial is to develop a health delivery system that effectively manages hypertension at primary care level.

Hypothesis: The development of an integrated management approach will be effective in managing hypertension at all levels among hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40 years or over visiting the selected IMS centre with known hypertension or with consistently elevated BP on two separate visits (mean of last two of three measurements of systolic pressure ≥140 mm Hg or mean diastolic pressure ≥90 mm Hg) or already receiving treatment will be eligible for inclusion in the study.

Exclusion Criteria:

* Those patients who require intensive care unit or coronary care unit admissions, or are diagnosed to have cognitive impairment, are agitated due to severe pain, non-resident of Karachi, or having language barrier will be excluded from the study.
* A screening form will be designed for the collection of the above mentioned information. The rationale of excluding all the participants with above mentioned condition is that the participants having these health concerns will either not be able to respond to our questionnaire or their presence may confound our results.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
At least an absolute 20% point greater proportion of participants in the intervention group achieving blood pressure targets ( SBP <140 mmHg and DBP < 90mmHg) | 6 months

SECONDARY OUTCOMES:
Adherence to life style modification | 6 months
  Adherence to life style modification (exercise, diet, medication) by the patients: This will be assessed through self-report, anthropometric and blood pressure measurement and empty blister count at the follow up visits.
Adherence by physicians to hypertension management guidelines | 6 months
  Adherence by physicians to hypertension management guidelines: assessed through monthly audits conducted by the research medical officer.
Cost-Effectiveness | 6 months
  Cost-Effectiveness: cost of medication (self-report by patient), cost of physician visit (clinic data) etc.
Patient Satisfaction | 6 months
  Patient Satisfaction: This would be assessed through PSQ-18.

CONTACTS AND LOCATIONS:
Overall Officials: Waris Qidwai, Principal Investigator — Aga Khan University
Locations (1):
- The Integrated Medical Services Clinics (IMS), Karachi, Sindh, Pakistan